CLINICAL TRIAL: NCT07092345
Title: An Adaptive Intervention to Increase Engagement to Community-based Care After an ED Admission: For Youth at Risk for Suicide and Self-injurious Behavior
Brief Title: An Adaptive Intervention to Increase Engagement to Community-Based Care After an ED Admission
Acronym: ED_SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2037770; K23MH136332 (NIH)
Record Dates: First submitted 2025-03-17; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Suicidal and Self-injurious Behavior; Linkage to Care
Keywords: suicidality; self-injurious behavior; adaptive intervention; emergency department; caregivers; youth
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Emergencies

STUDY DESIGN:
Intervention Model Description: Adaptive intervention via Sequential Multiple Assignment Randomized Trial (SMART) design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Psychosocial (Experimental): Digitally delivered psychosocial
  Interventions: Behavioral: adaptive intervention
- Psychosocial with text messages (Experimental): Digitally delivered psychosocial with text messages
  Interventions: Behavioral: adaptive intervention
- Psychosocial with text messages and family navigator (Experimental): Digitally delivered psychosocial with text messages and human family navigator
  Interventions: Behavioral: adaptive intervention

INTERVENTIONS:
Behavioral: adaptive intervention — We will utilize an adaptive interventions via Sequential Multiple Assignment Randomized Trial (SMART) design provide a tailored, stepped-care approach for the type, intensity, and dose of treatment, thus, providing the most intensive care to only those who need it, particularly treatment non-response. First, youth and caregivers (dyads) will be randomized to receive 1st-stage interventions in the ED, either the digital psychosocial-only (PS) condition or the psychosocial with digital health communication (PS+text) condition. If identified as non-response at 2-weeks, then dyads will be re-randomized to 2nd-stage intervention(s). Specifically, the PS condition non-responders will be re-randomized to the PS+text condition or the PS+text+FN condition. The 1st-stage PS+text condition non-responders will receive the PS+text+FN condition only.

SUMMARY:
The goal of this study is to develop a feasible brief, family-based adaptive intervention, via SMART design, for youth with suicidal and non-suicidal self-injurious behavior (SSIB) to increase community-based mental health (MH) care attendance and reduce SSIB risk post emergency department (ED) admission. The intervention will focus to increase understanding on youth MH literacy, MH communication, and MH engagement. Integrating an adaptive intervention via a SMART design in the ED could address subsequent barriers to youth obtaining appropriate level of community-based MH care and therefore reduce ED readmissions.

DETAILED DESCRIPTION:
This adaptive intervention allows for two stages of randomization to address treatment non-response. First, youth and caregivers (dyads) will be randomized to receive 1st-stage interventions in the ED, either the digital psychosocial-only condition or the psychosocial with digital health communication via text messages condition. If after two weeks, youth are identified as non-response, then dyads will be re-randomized to 2nd-stage intervention(s) that will include the use of a family navigation model.

ELIGIBILITY:
Inclusion Criteria:

* Youth 8 to 17 years
* Youth presenting to the ED with suicide and self-injurious behavior
* Youth living at home with at least one legal guardian/caregiver

Exclusion Criteria:

* Youth presenting to the ED with psychosis, sexual assault, child abuse
* Youth in police custody,
* Youth with an active investigation with the department of child and youth services (DCYF)
* Youth unable to assent due to severity of illness or developmental disabilities,
* Youth who cannot communicate in English or Spanish,
* Youth without a caregiver/legal guardian who can provide consent

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | 3-month & 6-month follow-up assessments
  Recruitment rate (% of ppl who agree to be in the study), Study completion (% of ppl who complete entire study)
Child and Adolescent Service Assessment (CASA) | 3-month and 6-month follow-up assessments
  Youth Attendance to Community-based Mental Health Care. CASA question and caregiver report of youth attendance in behavioral health care/community-based mental health services (yes or no) after discharge from emergency department admission.
Intervention Acceptability | 3-month and 6-month follow-up assessments
  Client Satisfaction Questionnaire. An 8-item questionnaire that provides (positive & negative) feedback from user opinion. Higher scores = greater satisfaction with intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasbro Children's Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Cancilliere MK, Ramanathan A, Hoffman P, Jencks J, Spirito A, Donise K. Characteristics of a Pediatric Emergency Psychiatric Telephone Triage Service. Pediatr Emerg Care. 2022 Oct 1;38(10):494-501. doi: 10.1097/PEC.0000000000002831. Epub 2022 Aug 18. PMID 35981327
- [Background] Spirito A, Simon V, Cancilliere MK, Stein R, Norcott C, Loranger K, Prinstein MJ. Outpatient psychotherapy practice with adolescents following psychiatric hospitalization for suicide ideation or a suicide attempt. Clin Child Psychol Psychiatry. 2011 Jan;16(1):53-64. doi: 10.1177/1359104509352893. Epub 2010 Apr 19. PMID 20404070
- [Background] Cancilliere MK, Donise K. A Comparison of Acute Mental Health Presentations to Emergency Services Before and During the COVID-19 Pandemic. R I Med J (2013). 2022 May 2;105(4):9-15. PMID 35476729
- [Background] Cancilliere MK, Guthrie KM, Donise K, Lin T, Orchowski L, Spirito A. Development of an Emergency Department Family Navigator and Text Message Intervention for Caregivers to Reduce Youth Risk of Suicide and Self-injurious Behavior. R I Med J (2013). 2024 Aug 1;107(8):28-38. PMID 39058987